CLINICAL TRIAL: NCT06582706
Title: Nicotinic Acid for the Treatment of Alzheimer's Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Principal Investigator, Jared Brosch, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23519
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-01

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: This study is a randomized, placebo controlled, blinded trial that includes a single intervention arm. The intervention is extended release niacin 500mg. The control/placebo group will use microcrystalline cellulose tablets.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The size and shape of the placebo pill will be chosen to most closely match the other treatment tablets. The drugs will be placed into identical bottles and will be labeled with a unique identifier and stored in a locked, temperature monitored room. Randomization instructions from RedCap will designate a participant and their assigned uniquely identified bottle which will be given to them at randomization with instructions. At the 30-day visit a pill count will be undertaken to reinforce compliance. The bottle and any remaining pills will be collected at the end of the study and compliance will be assessed. All pill counts and pill instructions will be given by a separate study coordinator (due to inability to have a perfectly matching placebo) so that primary study coordinator and principal investigator remain blinded throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Extended -Release Niacin (Experimental): 500 mg daily
  Interventions: Drug: Extended Release Niacin
- Placebo (Placebo Comparator): Microcrystalline cellulose tablets
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Placebo Comparator — a readily available inert placebo will be used
  Other Names: microcrystalline cellulose tablets
  Arms: Placebo
Drug: Extended Release Niacin — 500 mg
  Arms: Extended -Release Niacin

SUMMARY:
Increased dietary intake of niacin is correlated with reduced risk of Alzheimer's Disease and age-associated cognitive decline. The goal of this study is to collect data on the penetration of commercially available, FDA approved, extended-release niacin into the spinal fluid. One dose of 500 mg nicotinic acid will be used (in addition to placebo) to build a dose response curve for this compound in human cerebrospinal fluid. This objective will demonstrate target engagement of HCAR2 in the central nervous system, after oral treatment with niacin. The primary endpoints are to show increased nicotinic acid levels in blood and cerebrospinal fluid. A secondary endpoint is to collect safety and tolerability data of niacin in this particular population.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a highly prevalent neurodegenerative disorder with several modestly effective therapies. Interestingly, increased dietary intake of niacin is correlated with reduced risk of AD and age-associated cognitive decline. Niacin/nicotinic acid is obtained principally through diet and can cross the blood brain barrier. Overall data support that niacin can be beneficial at mid/late AD stages limiting both amyloid and tau pathologies. Niacin formulations are currently being tested in clinical trials for Parkinson's disease and glioblastoma (NCT04677049 and NCT03808961) and are FDA-approved to treat dyslipidemia and its safety profile established in the general population. Thus, we propose a phase 2a clinical trial targeting microglia response by repurposing an FDA-approved formulation of niacin. This study (randomized, placebo controlled, blinded) includes a single intervention arm. The intervention is extended release niacin 500mg. The control/placebo group will use microcrystalline cellulose tablets. The size and shape of the placebo pill will be chosen to most closely match the other treatment tablets.

Following randomization, participants will receive their uniquely assigned drug bottle with instructions. At the 30-day visit a pill count will be undertaken to reinforce compliance. The bottle and any remaining pills will be collected at the end of the study and compliance will be assessed. All pill counts and pill instructions will be given by a separate study coordinator (due to inability to have a perfectly matching placebo) so that primary study coordinator and principal investigator remain blinded throughout the study. A compliance rate of 85% or better (approximately 9 missed doses over the 60 day period) is expected. Participants and study partners will be instructed to take their dose at the same time every morning. The pills should not be distributed into pill containers and retained within the study drug bottle. If a dose is missed and it is less than 12 hours from the missed dose, it should be taken immediately, otherwise it will be considered a "missed dose". Missing more than 15% of doses will lead to an early termination from the study. Pill count is completed at the interim visit.

At the screening visit patients will be appropriately screened for inclusion/exclusion criteria. Contraindicated medications will be reviewed. Integrity of the relationship between the participant and study partner will be ascertained; EKG and basic laboratory studies including hepatic function testing and coagulation studies will be reviewed. Physical and Neurologic examination will take place. All criteria will be reviewed, and the inclusion/exclusion criteria will be reviewed again at randomization. At randomization the participant will undergo additional cognitive and functional assessments, additional blood work will be drawn, and a lumbar puncture will be performed to obtain approximately 20 ml of cerebrospinal fluid (CSF). At week 4 a safety assessment and blood draw will take place along with pill counts and recording of adverse events (AEs). The final visit at week 8 will mirror the randomization visit with blood work, CSF collection, and cognitive and functional assessments.

ELIGIBILITY:
Inclusion Criteria:

Age 60-85 males or females

Clinically have a diagnosis of Alzheimer's disease in the mild-moderate dementia range Mini Mental Status Examination (MMSE) between 14-24 inclusive

Must be on a stable dose (30 days minimum) of a cholinesterase inhibitor and/or memantine (or absence thereof)

Have a reliable co-participant who has at least 3 days of face-to-face contact per week with the patient and ensures medical compliance with the study drug.

Neuroimaging (MRI or CT scan of the brain) should be available within 1 year of screening

Exclusion Criteria:

Any contraindication to clinical lumbar puncture including increased intracranial pressure, posterior fossa mass, bleeding diathesis, use of antiplatelet medications other than aspirin, use of any anticoagulant

Severe cerebrovascular disease

History of large territory stroke

Allergy or sensitivity to B-vitamins or nicotinic acid

History of elevated liver function tests (ALT/AST > 2x the upper limit of normal) or known liver disease

Current consumption of Vitamin B3 (any form, including nicotinic acid) - including multivitamins and energy drinks. Participants taking a supplement containing Niacin must washout for 4 weeks prior to screening to participate.

Renal impairment of Stage 2 or greater

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in nicotinic acid levels in blood and CSF | Baseline and 60 day visit
  Target engagement of HCAR2 in the CNS after treatment with niacin

SECONDARY OUTCOMES:
Number of participants with treatment related adverse events | Baseline to 60 day visit
  Adverse events will be collected throughout the study. Adverse events deemed related to nicotinic acid will be delineated from procedural based adverse events by the PI.

CONTACTS AND LOCATIONS:
Overall Officials: Jared R Brosch, MD, Principal Investigator — Indiana University
Locations (1):
- IU Health Neuroscience Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No